CLINICAL TRIAL: NCT03299868
Title: Comparison of Safety, Efficacy, and Patient-perceived Satisfaction Between Initial Routine Peripherally Inserted Central Catheters Insertion and General Intravenous Access in Terminally Ill Cancer Patients: A Randomized Phase II Study
Brief Title: Comparison Between Initial Routine PICC and General IV Access in Terminally Ill Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kwonoh Park, MD phD, Professor, clinical research, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEPTIC II
Record Dates: First submitted 2017-09-19; First posted 2017-10-03 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Peripherally Inserted Central Catheter; Intravenous Access
Keywords: Peripherally inserted central catheter; Terminally ill cancer patients; Palliative care
MeSH Terms: interventions — Catheterization, Peripheral

STUDY DESIGN:
Intervention Model Description: Prospective, Single institution, Open-label, Randomized, Phase 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine PICC group (Experimental): PICC is initially routine insertion at the time of admission of hospice-palliative care unit
  Interventions: Device: peripherally inserted central catheter (PICC)
- General IV group (Active Comparator): PICC is inserted if 3 or more times of IV insertion trial per day is required for IV access
  Interventions: Device: peripherally inserted central catheter (PICC)

INTERVENTIONS:
Device: peripherally inserted central catheter (PICC) — comparisons of the safety, efficacy, and patient-perceived satisfaction between the initially routine PICC insertion group (routine PICC group) and general IV access group (general IV group)

SUMMARY:
To establish the IV access strategy for terminally ill cancer patients, using comparisons of the safety, efficacy, and patient-perceived satisfaction between the initially routine PICC insertion group (routine PICC group) and general IV access group (optional PICC group).

DETAILED DESCRIPTION:
Reliable intravenous (IV) access is an important issue in terminally ill cancer patients, however, they have limited or no peripheral venous access due to edema or long period of IV therapy. Thus, intravenous access has been provided by Central venous catheter (CVC).

There are some options for applying CVC in cancer patients; subclavian venous catheter (SVC), chemo-port (CP), and the peripherally inserted central catheter (PICC).

When considering the characteristics of terminally ill cancer patients, such as poor general condition and a limited period of survival, PICC could be a safe and effective method for intravenous access.

There are two previous studies concerned about PICC study in terminally ill cancer patients. They showed that PICC might be overall safe and efficient in terminally ill cancer patients. However, these studies did not evaluate superiority of PICC insertion compared to no insertion and the appropriate time for PICC insertion due to limitation of their design, such as retrospective or single-arm observational study. Thus, strategies of PICC insertion for IV access in terminally ill cancer patients have not been determined until now.

Considering the favorable results of PICC insertion in previous studies and limited survival time of terminally ill cancer patients, the investigator postulated that routine PICC insertion at the time of admission for terminal care would be effective for IV access.

Thus, the investigator assumed that initially routine PICC insertion would be non-inferior in maintenance success rate / and complication rate compared to general IV access. In addition, it would be superior in patient-perceived satisfaction. The inveistigator will undertake a randomized phase II study to confirm the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients with histologically or cytologically confirmed malignancy and fulfilled all of the following conditions
2. Patients with expected survival time of 3 months or less due to a progressive disease without additional anticancer treatment. (However, palliative radiation treatment for symptom control is allowed.)
3. Patients who need the IV access route continuously for hydration or medication.
4. Age18 or older
5. Signed and dated informed consent of document indicating that the patient (or legally acceptable representative) has been informed about all pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

1. Patients who showed severe coagulopathy such as thrombocytopenia (Platelet count ≤ 20,000/mm2) or international normalized ratio (INR) prolongation (≥2.0 ) in spite of treatment
2. Patients who have an evidence of current sepsis (bacteremia or fungemia)

   1. 'current' means bacteremia/fungemia without eradication on follow-up peripheral blood culture
   2. patients with persistent fever (bacteremia or fungemia cannot be ruled out)
3. Patients who is impracticable to PICC insertion due to uncontrolled behavioral disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
IV access maintenance success rate | From date of enrollment until death or discharge/transfer, assess up to 2 years
  rate of successful PICC maintenance until death or discharge/transfer

SECONDARY OUTCOMES:
PICC related complication rate | From date of enrollment until death or discharge/transfer, assess up to 2 years
  rate of any complication which is related with PICC
PICC premature removal rate | From date of enrollment until date of PICC removal, assess up to 2 years
  rate of premature removal such as self-removal or CRBSI before death or discharge
PICC life span | From date of enrollment until death or discharge/transfer, assess up to 2 years
  median survival of PICC
patient perceived procedure-related distress | 5th day after procedure
  procedure-related distress during insertion of PICC
patient perceived comfort and convenience assessed by a newly developed question in this study | 3th to 7th day after enrollment
  patient perceived comfort and convenience ("How do participants feel comfort and convenience about the IV access?" at 3th - 7th days after enrollment
colonization of microbiology in PICC | at the time of PICC removal, assess up to 2 years
  Investigator evaluate the colonization of PICC using tip culture at the time of removal

CONTACTS AND LOCATIONS:
Overall Officials: Kwonoh Park, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cleeland CS. Cancer-related symptoms. Semin Radiat Oncol. 2000 Jul;10(3):175-90. doi: 10.1053/srao.2000.6590. PMID 11034629
- [Result] Bruera E, Sala R, Rico MA, Moyano J, Centeno C, Willey J, Palmer JL. Effects of parenteral hydration in terminally ill cancer patients: a preliminary study. J Clin Oncol. 2005 Apr 1;23(10):2366-71. doi: 10.1200/JCO.2005.04.069. PMID 15800328
- [Result] Mercadante S, Ferrera P, Girelli D, Casuccio A. Patients' and relatives' perceptions about intravenous and subcutaneous hydration. J Pain Symptom Manage. 2005 Oct;30(4):354-8. doi: 10.1016/j.jpainsymman.2005.04.004. PMID 16256899
- [Result] Lam S, Scannell R, Roessler D, Smith MA. Peripherally inserted central catheters in an acute-care hospital. Arch Intern Med. 1994 Aug 22;154(16):1833-7. PMID 8053751
- [Result] Ng PK, Ault MJ, Ellrodt AG, Maldonado L. Peripherally inserted central catheters in general medicine. Mayo Clin Proc. 1997 Mar;72(3):225-33. doi: 10.4065/72.3.225. PMID 9070197
- [Result] Raad I, Davis S, Becker M, Hohn D, Houston D, Umphrey J, Bodey GP. Low infection rate and long durability of nontunneled silastic catheters. A safe and cost-effective alternative for long-term venous access. Arch Intern Med. 1993 Aug 9;153(15):1791-6. PMID 8392831
- [Result] Smith JR, Friedell ML, Cheatham ML, Martin SP, Cohen MJ, Horowitz JD. Peripherally inserted central catheters revisited. Am J Surg. 1998 Aug;176(2):208-11. doi: 10.1016/s0002-9610(98)00121-4. PMID 9737634
- [Result] Park K, Jun HJ, Oh SY. Safety, efficacy, and patient-perceived satisfaction of peripherally inserted central catheters in terminally ill cancer patients: a prospective multicenter observational study. Support Care Cancer. 2016 Dec;24(12):4987-4992. doi: 10.1007/s00520-016-3360-6. Epub 2016 Jul 26. PMID 27460015